CLINICAL TRIAL: NCT06819917
Title: Prospective Sample Collection Study for Discovery and Evaluation of Novel Blood Based Biomarkers for Assessment of Hepatic Fibrosis
Brief Title: Identification of Liver Fibrosis Biomarkers
Status: Not yet recruiting | Type: Observational
Sponsor: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RD006521
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Non-alcoholic Fatty Liver; Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Identification of liver fibrosis biomarkers — Patients will be recruited in the study using 2 different approaches. The first is patients who are referred to clinical centers as part of an existing assessment where a decision to perform a liver biopsy has been made (routine biopsy). This decision can be based on standard liver function tests AST, ALT, FIB-4 (performed up to 8 months before biopsy), fibroscan (performed up to 6 months before biopsy) or other factors.
  In addition, patients F0-F2 who underwent a biopsy within the last 6 months but at least 1 month ago, can be recalled to join the study. If patients agree to participate in the study, they will be recalled to the site for a blood draw and ultrasound scan.

SUMMARY:
Chronic liver disease (CLD) is a major cause of global mortality and morbidity . CLD patients are at an increased risk of developing liver fibrosis (formation of scar tissue), cirrhosis and liver failure and are at significant risk to develop primary liver cancer. Non-alcoholic fatty liver disease (NAFLD) represents a major risk for CLD and it is becoming the most common chronic liver condition with an estimated 25% global prevalence. Progression to non-alcoholic steatohepatitis (NASH) occurs in approx. 1 of 5 NAFLD patients and due to the rapidly rising etiology of end-stage liver disease, is currently the second most common etiology of hepatocellular carcinoma (HCC) requiring liver transplantation. Liver biopsy, currently the gold-standard for grading disease activity and staging fibrosis, is invasive, costly and at risk for sampling error. Due to the number of patients diagnosed with fibrosis and since fibrosis stage is prognostic of mortality and drives patient management, it is important to develop noninvasive yet accurate diagnostic tools that can identify fibrosis stage. The purpose of this study is to obtain a panel of clinically well characterized blood specimens to identify novel biomarkers to be used as an aid in diagnosis to assess the stage of clinically significant hepatic fibrosis in patients with signs or symptoms of NAFLD (NAFL/NASH). In addition, quantitative ultrasound (QUS) based approaches combined with artificial intelligence (AI) algorithms will be explored for assessing the stage of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for biopsy (or F0-F2 patients that underwent biopsy within the last 6 months but at least 1 month ago) suspected of having hepatic fibrosis due to NAFLD (NAFL/NASH) or patients with MASLD or MASH
* Any FIB-4 value available
* Any Fibroscan value available
* Written and signed informed consent present
* Patients aged ≥ 18 years to ≤ 75 years at the time of the blood draw
* Body Mass Index (BMI) ≤ 45 kg/m²

Exclusion Criteria:

* Vulnerable person: person deprived of liberty by a judicial or administrative decision and/or person under psychiatric care
* Self-reported pregnancy or lactating females
* Disease related to other etiologies, including alcoholic liver disease (alcoholic steatohepatitis), MetALD, specific etiology SLD (e.g. DILI or monogenic disease), cryptogenic SLD, viral hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis, human immunodeficiency virus, Wilson's disease, Hemochromatosis, alpha-1 antitrypsin deficiency
* Any type of carcinoma, unless it is at least 5 years in remission
* Prior liver transplant
* Evidence of any other unstable or, untreated clinically significant immunological, neoplastic, endocrine, haematological, gastrointestinal, neurological or psychiatric disorder. Medically controlled comorbidities can be allowed
* Self-reported alcohol consumption greater 30 g/day (males) 20 g/day (females)
* Recent myocardial infarction (within last 6 months)
* Inability to have a liver biopsy, or provide blood sample in a fasted status
* F0-F2 recalled patients with +/- 5% change in weight between the biopsy and study inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in the study using 2 different approaches. The first is patients who are referred to clinical centers as part of an existing assessment where a decision to perform a liver biopsy has been made. This decision can be based on standard liver function tests AST, ALT, FIB-4 , fibroscan or other factors.
  In addition, patients F0-F2 who underwent a biopsy within the last 6 months but at least 1 month ago, can be recalled to join the study. If patients agree to participate in the study, they will be recalled to the site for a blood draw and ultrasound scan (if patients consent for further use, to be performed latest 6 months after biopsy).
Sampling Method: Probability Sample
Enrollment: 575 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Identification of Significant Fibrosis (≥F2) | Through study completion, an average of 1 year.
  The study aims to identify significant liver fibrosis (stage F2 or higher) through various biomarkers. This involves the comparison of biomarkers to biopsy results to determine their predictive value .
Identification of Advanced Fibrosis (≥F3) | Through study completion, an average of 1 year.
  he study aims to identify advanced liver fibrosis (stage F3 or higher) through various biomarkers. The assessment will determine the predictive value of these biomarkers for advanced stages of fibrosis (F3-F4)

SECONDARY OUTCOMES:
Performance of Biomarkers in Clinically Relevant Subpopulations | Through study completion, an average of 1 year.
  Exploratory analysis to evaluate the performance of identified biomarkers within specific patient sub-groups. This aims to understand the variability and reliability of biomarkers across different demographics and clinical characteristics.
Evaluation of Biomarker Panels | Through study completion, an average of 1 year.
  This measure involves evaluating individual or combined biomarkers identified through literature review, pathway analysis, and experimental programs using a panel of well-characterized blood specimens (serum, plasma, whole blood, and buffy coat).

IPD SHARING:
Plan to Share IPD: Undecided